CLINICAL TRIAL: NCT02158819
Title: A Prospective, Randomised Pilot Study to Compare Health Economic Outcomes Using a Patient-matched Cutting Guide Versus Standard Instrumentation in Total Knee Arthroplasty.
Brief Title: Visionaire Health Economics Study Comparing Economic Outcomes Between Visionaire and Standard Instrumentation
Acronym: VISHE13
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VISHE.13
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Visionaire; Health Economics; Degenerative arthritis; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TKA with standard instrumentation (No Intervention): This arm consists of the Genesis II Total knee implant system or the Legion Primary total knee system with standard instrumentation
- Total knee arthroplasty with Visionaire (Active Comparator): This arm will consist of the Genesis II Total Knee Implant System or Legion Primary Total Knee System with the Visionaire patient-matched instrumentation
  Interventions: Device: Total knee arthroplasty with Visionaire

INTERVENTIONS:
Device: Total knee arthroplasty with Visionaire — Patient Specific Instrumentation
  Arms: Total knee arthroplasty with Visionaire

SUMMARY:
The purpose and primary objective of this study is to compare health economic outcomes between the use of a patient-matched cutting guide (Visionaire) versus the use of standard instrumentation in Total Knee Arthroplasty(TKA). Data will be collected pre-operatively, intra-operatively and post operatively up until and including the six week post-operative assessment. The secondary objectives of the study are to compare safety and early readmission rates between the two techniques. The study hypothesis is that there is no difference in the cost of the episode of care from hospital admission to discharge, including pre-operative radiology costs and cost of resources, with the Visonaire patient-matched cutting guide compared to standard instrumentation.

DETAILED DESCRIPTION:
This is a prospective, randomised pilot study comparing the health economic outcomes between TKA using standard instrumentation and TKA using a patient-matched cutting guide. The primary indication for this study is degenerative arthritis of the knee requiring unilateral primary total knee arthroplasty. Patients requiring TKA who are eligible and have consented to participate will be randomised to TKA with The Genesis II™ Total Knee Implant System or the Legion™ Primary Total Knee System using either Visionaire™ patient-matched cutting guides or standard instrumentation. The study will recruit for 1 year and patients will have a final follow up at the six week post-operative assessment.

The primary objective of this study will evaluate the cost of the episode of care from hospital admission to discharge. This will include pre-operative costs, anesthetic costs, operative and theatre costs, costs of instruments and resources. The study will also measure length of stay as well as blood transfusion requirements. The secondary objectives of this study are to compare the safety and early readmission rates between the two techniques, by measuring the complication rates intra-operatively and post-operatively as well as the number of patients readmitted to hospital prior to the six week post-operative assessment.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative arthritis of the knee requiring unilateral primary Total Knee Arthroplasty in subjects for whom the use of patient-matched cutting guides or standard instrumentation are, in the surgeon's opinion, clinically appropriate and acceptable forms of treatment;
* Patient is of legal age to consent and is skeletally mature;
* The patient is able to fully understand the purpose of the trial, and his/her role as a participant in the study
* The patient consents to his/her inclusion in the study after the nature, scope and possible consequences of the study have been explained in an understandable form.

Exclusion Criteria:

* Patient is known to have poor bone stock making a Total Knee Arthroplasty unjustifiable.
* Patient is immuno-suppressed.
* Patient has physical, emotional or neurological conditions that would compromise the subject's compliance with postoperative rehabilitation and follow-up.
* Patient is pregnant or may become pregnant during the course of the study, or is lactating.
* Patient has a history of prior ipsilateral major knee surgery (e.g. arthroplasty, high tibial osteotomy, or tibial plateau fracture). Minor prior procedures such as Anterior Cruciate Ligament repair, meniscectomy, or arthroscopy are not excluded.
* Patient has active, localized or systemic infection.
* Patient is severely overweight (BMI >40).
* Patient is a prisoner.
* Patient has a significant MRI (magnetic resonance imaging) exclusion or contraindication.
* Patient has had a total joint arthroplasty of the contralateral limb in the last 12 months.
* Patient presently identified with future need for bilateral TKA within the next twenty-four months.
* Patient has a known or suspected hypersensitivity/allergy to foreign materials contained in the implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Cost of the episode of care from admission to hospital to discharge | up to 1 week
  The cost of the episode of care from admission to hospital to discharge , including pre-operative radiology costs and costs associated with Visionaire and will incorporate the costs of time, number of instruments utilised, blood transfusion requirements, length of stay and pre-operative xray and MRI costs.

SECONDARY OUTCOMES:
Percentage of patients that experience short term complications and/or early readmissions | up to 6 weeks
  Percentage of patients experiencing intra-operative complications, post operative complications, post discharge complications or readmissions prior to the 6 week post-operative assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Baker, Principal Investigator — Private Practice; Lieth Stewart, Principal Investigator — Life Claremont Hospital; Willem Tollig, Principal Investigator — Pretoria East Hospital; Michael Barrow, Principal Investigator — Sunninghill Hospital; Dan Potgieter, Principal Investigator — Life Bay View Hospital
Locations (5):
- South Africa (5):
  - Life Bay View Hospital, Mossel Bay, Cape Town
  - Sunninghill Hospital, Johannesburg, Gauteng
  - Pretoria East Hospital, Pretoria, Gauteng
  - Private Practice, Durban, KwaZulu-Natal
  - Life Claremont Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No